CLINICAL TRIAL: NCT02737241
Title: Randomized Clinical Trial Comparing Low Power (50W) Holmium Laser Enucleation of the Prostate (HoLEP) Versus High Power (100W) HoLEP
Brief Title: HoLEP (50W) vs. HoLEP (100W) for Treatment of BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mans 26-11-2015
Record Dates: First submitted 2016-03-27; First posted 2016-04-13 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Prostatic Hyperplasia
Keywords: Prostate; Laser; Enucleation
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LP-HoLEP (Active Comparator): Low power Holmium laser enucleation of the prostate
  Interventions: Procedure: Low power Holmium laser enucleation of the prostate
- HP-HoLEP (Active Comparator): High power Holmium laser enucleation of the prostate
  Interventions: Procedure: High power Holmium laser enucleation of the prostate

INTERVENTIONS:
Procedure: Low power Holmium laser enucleation of the prostate — HoLEP entails dissection of the whole median and lateral prostatic lobes off the surgical capsule via a retrograde approach starting at the apex. The enucleated lobes were pushed to the bladder followed by hemostasis of the prostate bed then intravesical morcellation of the enucleated adenoma. The procedure entails power setting of 50W holmium laser energy.
  Arms: LP-HoLEP
Procedure: High power Holmium laser enucleation of the prostate — HoLEP entails dissection of the whole median and lateral prostatic lobes off the surgical capsule via a retrograde approach starting at the apex. The enucleated lobes were pushed to the bladder followed by hemostasis of the prostate bed then intravesical morcellation of the enucleated adenoma. The procedure entails power setting of 100W holmium laser energy.
  Arms: HP-HoLEP

SUMMARY:
HoLEP (Holmium laser enucleation of the prostate) entails dissection of the whole median and lateral prostatic lobes off the surgical capsule via a retrograde approach starting at the apex. The enucleated lobes were pushed to the bladder followed by hemostasis of the prostate bed then intravesical morcellation of the enucleated adenoma.

The investigators are going to compare safety and efficacy of low power; LP-HoLEP vs. high power; HP-HoLEP in treatment of infra-vesical obstruction secondary to BPH (Benign prostate Hyperplasia).

DETAILED DESCRIPTION:
Introduction

Benign prostatic hyperplasia (BPH) is a pathologic process that contributes to, but is not the sole cause of, lower urinary tract symptoms (LUTS) in aging men.

The decision to intervene is frequently used as an end point after failure of different medical therapies. These medications are able to delay this point. Failed medical treatment either due to refractory LUTS or in patients who are not willing to make a lifetime commitment to medical therapy represents one indication to intervene.

Urine retention secondary to BPH with failed voiding trial without catheter is an indication for intervention in healthy individuals as well as recurrent hematuria, secondary vesical stones and recurrent urinary tract infection. Renal deterioration secondary to BPH is an indication of intervention after proper evaluation of the bladder function.

For years, surgical treatment for BPH was transurethral resection of the prostate (TURP) for small to moderate sized prostate and open prostatectomy (OP) for markedly enlarged one.

Laser prostatectomy was introduced as a less invasive modality for treatment of BPH overcoming the disadvantages and limitations of the traditional standard TURP and OP. It seems to be advantageous as it is less invasive than OP. Furthermore, using physiological saline as an irrigant, with higher safety profile in morbid patients who have to be on anticoagulants or antiplatelet during surgery. It is used to tackle larger prostate glands beyond the limits of TURP. It is not infrequent to be done as day surgery with shortened catheterization time.

Eventually it seems to be cost effective, however the remaining concern as in all minimally invasive surgeries (MIS) is the durability and reoperation rates. Despite the significant advantages known with laser prostatectomy techniques particularly HoLEP, adoption of these procedures in urologic community is limited and one of the causes is the high initial cost investment for laser capital equipment.

HoLEP entails dissection of the whole median and lateral prostatic lobes off the surgical capsule via a retrograde approach starting at the apex. The enucleated lobes were pushed to the bladder followed by hemostasis of the prostate bed then intravesical morcellation of the enucleated adenoma.

Over the past 15 years, different technical modifications have come out to the procedure. However all the current reports use 100 watt laser power (High power HoLEP: HP-HoLEP) for the laser assisted enucleation technique.

Khan et al 2015, reported on the feasibility of using low power (LP-HoLEP) for safe and effective HoLEP. The authors cut significantly on the initial cost of laser capital equipment. They used 50-watt holmium laser machine to accomplish the enucleation procedure with reasonable efficacy. Nevertheless, there are no randomized studies assessing safety, efficacy and cost saving associated with LP-HoLEP.

Aim of the Work

This study aims to compare safety and efficacy of LP-HoLEP vs HP-HoLEP in treatment of infra-vesical obstruction secondary to BPH.

Patients and Methods

Study design: Randomized Controlled Trial (RCT)

Study population:

BPH surgical candidates presented to the outpatient clinic of the prostate unit in the urology department (Urology & nephrology center, Mansoura University) will be assessed to evaluate if these patients are eligible to the study inclusion criteria.

BPH surgical candidates are patients presented with LUTS secondary to BOO (bladder outlet obstruction) due to BPH who failed medical treatment, IPSS (international prostate symptom score) score >15, peak urinary flow rate (Qmax) <15 ml/sec, recurrent attacks of urine retention with failed trial voiding, patients with hematuria of prostatic origin with failed medical treatment and patients with vesical stone secondary to BPH.

Preoperative work up:

All patients will be thoroughly evaluated by medical history and physical exam, digital rectal exam (DRE), prostate specific antigen (PSA), urinalysis and urine culture, international index of prostate symptom score (IPSS), transrectal ultrasound (TRUS) measurement of prostatic volume and biopsy whenever indicated, measurement of post-void residual assessment (PVR), and maximum urinary flow rate (Qmax). Patients with positive urine culture will be treated accordingly.

Randomization:

Patients will be randomly assigned to the study groups on the day of the surgery after signing the informed consent for participation in the study. The randomization process will be performed using computer-generated random tables in a 1:1 ratio. A stratified-blocked randomization across two strata derived from predetermined size grouping (40-80 ml and more than 80 ml) and two strata derived from preoperative indication (catheterized and non-catheterized) were done. This method ensures parity among the two treatment groups. In each stratum, given two possible block lengths of four and eight respectively, with a random number generator giving numbers uniformly distributed between 0 and 1, the investigators selected a block length of four for random numbers lower than 0.5 or a block length of eight otherwise. Variation of the block sizes prevented the surgeon from guessing what the next treatment will be; it makes it difficult (although not impossible) to break the treatment code.

Eligible patients will be randomized into one of two groups:

Group 1 (50 patients): Patients will be managed with HP-HoLEP. Group 2 (50 patients): Patients will be managed with LP-HoLEP.

Procedure:

In case of coexisting urinary bladder stone, Holmium laser cystolithotripsy will be done first.

Laser setting:

* HP-HoLEP: (Energy=2 Joule, Rate=50 Hertz) for adenoma enucleation & reduced to (Energy=1.5, Rate=30) for apical dissection & hemostasis.
* LP-HoLEP: (Energy=2 Joule, Rate=25) throughout the whole procedure.

Surgical Technique:

HoLEP can be divided into four phases: inspection, enucleation, hemostasis and morcellation. Briefly, a plane was created between the adenoma and the surgical capsule early after the first incision of the gland from the bladder neck to the level of the verumontanum. The gland was enucleated in two or three lobes depending on the anatomy and the prominence of the grooves on either side of the middle lobe.

The Two-lobe technique starts with a 5- or 7-O'clock incision in a groove between the median lobe and one lateral lobe (the deeper groove) with enucleation of one lateral lobe, followed by the median and the remaining lateral lobe as a single unit.

The three-lobe technique involves a 5- and 7- O'clock incisions with enucleation of the median lobe and subsequent enucleation of one lateral lobe followed by the other lateral lobe.

If bleeding is encountered, the laser fiber can be defocused slightly from the bleeding point to achieve hemostasis.

Furosemide (20 mg/hour, intravenously) is administered after one hour of surgery, to correct for any fluid absorption and to enhance urine flow. After hemostasis, the morcellator is introduced and the prostatic lobes are morcellated and removed.

Follow-up:

Patients will be seen in follow-up at 2-4 weeks, 4 months, and 12 months.

Validated questionnaires will be utilized to assess the patients' sexual function both at base line and at different follow-up visits. Different aspects of the sexual function will be analyzed.

In patients who may have no symptomatic improvement after the procedure or who may have subsequent deterioration, cystoscopy will be performed to rule out the development of a urethral stricture or bladder neck contracture. Treatment will be planned accordingly for the present finding.

Outcome measures:

Primary outcomes:

The primary outcomes of this clinical trial will be operative outcome measures including:

Operative time; which is the time from insertion of the resectoscope till the time of catheterization, operative efficacy; which is the number or grams of the resected prostate tissue weight divided by operative time, enucleation efficacy (study endpoint); which is the number of grams of the resected prostate tissue divided by enucleation time, laser / prostate ratio; which is the amount of the joules of laser energy spent to remove one gram of the prostate tissue and the peri-procedure blood changes: Hg deficit, Hct deficit, Na changes.

Secondary outcomes:

These parameters include; time to catheter removal, duration of hospital stay and complications (intraoperative, early postoperative during first 30 days after the procedure, late postoperative).

Furthermore, urinary outcome measures (IPSS; international prostate symptoms score, QOL; quality of life, Q-max; peak flow rate, PVR; post voiding residual) and sexual outcome measures (Changes in the IIEF-15; international index of erectile function-15) will be depicted and compared.

Tertiary outcome:

The cumulative health resources related cost analysis of both procedures from a local institutional perspective (actual cost). Costs linked to the medical staff will not be included because they were assumed to be identical between the 2 groups, similarly routine clinic visits will not be included.

Participants' flow diagram (CONSORT CHART):

For each group, the numbers of participants who will be randomly assigned, receive intended treatment, and will be analyzed for the primary outcome. Losses and exclusions will be described in each group.

Sample size and statistical analysis:

In this study, the investigators will test the non-inferiority of LP-HoLEP to HP-HoLEP in accomplishing the transurethral enucleation procedure with comparable enucleation efficacy pertaining the advantages of lower cost and potential minimal postoperative dysuria.

Type 1 statistical error less than 5% and type 2 statistical error less than 20% were considered. Furthermore, based on previous report, enucleation efficacy using LP-HoLEP was reported as 0.68 + 0.4, 95%CI 0.61-0.75 gm/min (7) with an acceptable non-inferiority margin of 0.2gm/min was considered.

Considering the previous factors, a sample size of 100 patients (50 in each group) was estimated

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age ≥50 years
2. ASA (American society of anesthesiologists) score ≤3.
3. TRUS (transrectal ultrasound) estimated weight ≥40 grams.

Exclusion Criteria:

Patients who have any of the following were excluded:

1. Patient with neurological disorder which might affect bladder function as cerebrovascular stroke or Parkinson disease.
2. Active urinary tract infection.
3. Presence of bladder cancer (within the last 2 years).
4. Prostate cancer patients.
5. Patients with bleeding tendency, ongoing anticoagulants or antiplatelet medications
6. Previous prostate surgery

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Operative time (minutes) | one day
  Which is the time from insertion of the resectoscope till the time of catheterization
Operative efficacy (gm/minute) | one day
  Which is the number or grams of the resected prostate tissue weight divided by operative time
Enucleation efficacy (gm/minute) | one day
  Which is the number of grams of the resected prostate tissue divided by enucleation time

SECONDARY OUTCOMES:
dysuria score | 4 weeks
  Dysuria visual analogue scale will be used to assess postoperative dysuria at first postoperative visit
Maximum urine flow rate (ml/sec) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No